CLINICAL TRIAL: NCT04193657
Title: Toward a Comprehensive Supportive Care Intervention for Older or Frail Men With mCRPC
Acronym: TOPCOP2
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Prostate Cancer Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 19-5766
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Prostate Cancer; Older men; Supportive care; Frailty
MeSH Terms: conditions — Prostatic Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chemotherapy: 30 participants starting chemotherapy
  Interventions: Other: Daily and weekly triggered symptom monitoring
- Abiraterone: 20 participants starting Abiraterone
  Interventions: Other: Daily and weekly triggered symptom monitoring
- Enzalutamide: 20 participants starting Enzalutamide
  Interventions: Other: Daily and weekly triggered symptom monitoring
- Radium-223: 20 participants starting Radium-223
  Interventions: Other: Daily and weekly triggered symptom monitoring

INTERVENTIONS:
Other: Daily and weekly triggered symptom monitoring — Participants are invited to complete a daily questionnaire, a weekly questionnaire, and to track daily activity with an electronic activity tracker.
  Other Names: Daily Step count

SUMMARY:
1. Multicentre pilot study (n=90) which aims to study a prevalent population of elderly or frail patients with mCRPC whom are often excluded from clinical trial participation. (Data is sorely needed in this population)
2. The study aims to determine:

   1. if symptom monitoring (daily) is feasible using telephone or electronic means of communications in the elderly or frail patient with mCRPC
   2. The time course/pattern of symptoms important to quality of life for patients undergoing chemotherapy, abi/enza, or Radium 223
   3. If changes in physical activity (quantified by fitbit) predict for changes to ESAS in men undergoing treatment d) Qualitatively assess the supportive care needs of older/frail men with mCRPC

DETAILED DESCRIPTION:
Study Aim:

The previous multi-centre observational study (TOPCOP), funded by Prostate Cancer Canada, demonstrated important declines in multiple areas of quality of life, and fatigue and functional decline which were common issues that often limited further treatment. Emerging data from other settings demonstrate that (a) close monitoring of symptoms may reduce treatment toxicity and improve survival; (b) improving physical activity and targeting pain and sleep may improve fatigue and function. Whether these are feasible in the setting of older or frail men with mCRPC is unclear. Incorporating what the investigators have learned from TOPCOP and emerging supportive oncology literature, our main aim is to examine the emergence of key symptoms (fatigue, pain, insomnia) and explore whether reductions in daily physical activity are early indicators of toxicity over one treatment cycle (3-4 weeks) and therefore targetable in a subsequent intervention study.

Study Design:

This is a prospective multicentre observational study. The investigators will enroll English-speaking men with mCRPC who are either age 75 or older or age 60-74 and frail using (a) chemotherapy; (b) abiraterone or enzalutamide; (c) Radium.

Daily telephone-based brief symptom screening will be done with the Edmonton Symptom Assessment Scale (ESAS). Daily monitoring of physical activity (step counts) will be done with commercial smartphone apps or a Fitbit device. Moderate or higher symptoms (>3/10) on ESAS or a decrease in daily step count of 15% or more triggers more detailed telephone-based toxicity assessment and measures of pain, sleep, and fatigue as appropriate. The study duration is 3 weeks (1 cycle of chemotherapy) or 4 weeks (abiraterone/enzalutamide/radium). Qualitative interviews will be done to explore challenges with treatment tolerability and adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Starting either chemotherapy, Radium-223, Abiraterone or Enzalutamide or starting chemo > one year post CHAARTED
2. At least 65 years old
3. Able to provide written informed consent
4. Diagnosed with metastatic castrate resistant prostate cancer
5. Total Testosterone level 1.7nmol/L
6. Has a working smartphone OR is willing to use a study provided smartphone

Exclusion Criteria:

-

Min Age: 60 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer occurs in males only.
Study Population: 1. Unable to speak English fluently.
  2. Severe neuropsychiatric abnormalities.
  3. Limited life expectancy (<3 months) as estimated by the primary oncologist or seeing palliative care.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Daily monitoring with Edmonton Symptom Assessment Scale (ESAS) | 3-4 weeks
  Number of participants with treatment-related adverse events as measured by ESAS.Moderate or higher symptoms (>3/10) on ESAS triggers more detailed telephone-based toxicity assessment
Using a personal physical activity tracker step counts are monitored daily. | 3-4 weeks
  Number of participants with a decrease in daily step count of 15% or more that triggers more detailed telephone-based assessment.
Brief Pain Inventory-Short Form (BPI-SF) to measure pain severity | 3-4 weeks
  Number of participants with ESAS pain score greater than 3 that triggered BPI-SF. than 3
Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) to measure fatigue | 3-4 weeks
  Number of participants with ESAS fatigue score greater than 3 that triggered MFSI-SF.
Insomnia Severity Index (ISI) to measure treatment related insomnia | 3-4 weeks
  Number of participants with ESAS insomnia score greater than 3 that triggered ISI
Patient Health Questionnaire 9-item (PHQ-9) to measure treatment related depression | 3-4 weeks
  Number of participants with ESAS depression score greater than 3 that triggered PHQ-9.
Generalized Anxiety Disorder 7-item (GAD) to measure treatment related anxiety | 3-4 weeks
  Number of participants with ESAS anxiety score greater than 3 that triggered GAD

SECONDARY OUTCOMES:
Participants symptom experience by Qualitative interview | 30 minutes
  Participants in each treatment arm will be invited to participate in semi-structured one-time qualitative interviews after one cycle of treatment. The interview will focus on the symptom experience, impact on daily life, strategies used to manage symptoms, and suggestions for external support.
Study Completion Questionnaire to measure participant burden and satisfaction | 5 minutes
  Number of participants that experienced burden or satisfaction by the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided